CLINICAL TRIAL: NCT06514222
Title: Pain Control Following Impacted Mandibular Third Molar Surgery: A Comparison of the Effectiveness of Two Different Protocols
Brief Title: Pain Control Following Third Molar Surgery
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Kamis Gaballah, Program Director for MDS-Oral Surgery, Associate Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-23-03-25-01-S
Record Dates: First submitted 2024-07-08; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain; Impacted Third Molar Tooth
Keywords: Third molar surgery; Post Operative Pain; Paracetamol; Ibuprofen
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: A single-center, double-blind, parallel-group, randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluators responsible for data collection and analyses are blinded to the analgesic medication regime used by the patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study (Experimental): patient will receive 400mg ibuprofen and 1000mg Paracetamol at 4 hours in intervals for two days. With a total of 3 doses of ibuprofen and 3 doses of paracetamol per day
  Interventions: Drug: Paracetamol and Ibuprofen. The combination of the Paracetamol and Ibuprofen will be given together every 8 hours
- Control (Active Comparator): The patient will receive 400mg of ibuprofen plus 1000mg of Paracetamol simultaneously every 8 hours for two days.
  Interventions: Drug: Paracetamol and Ibuprofen. The combination of the Paracetamol and Ibuprofen will be given alternatively every four hours

INTERVENTIONS:
Drug: Paracetamol and Ibuprofen. The combination of the Paracetamol and Ibuprofen will be given together every 8 hours — Group 1- The patient will receive 400mg ibuprofen plus 1000mg Paracetamol simultaneously every 8 hours for two days.
  Arms: study
Drug: Paracetamol and Ibuprofen. The combination of the Paracetamol and Ibuprofen will be given alternatively every four hours — Group 2- The patient will receive 400mg ibuprofen and 1000mg Paracetamol at 4 hours in intervals for two days. With a total of 3 doses of ibuprofen and 3 doses of paracetamol per day
  Arms: Control

SUMMARY:
In this study, the investigators recruited patients undergoing surgical removal of impacted third molar teeth. Participants will be randomly divided into two groups Group 1: The patient will receive 400mg of ibuprofen plus 1000mg of Paracetamol simultaneously every 8 hours for two days.

Group 2- The patient will receive 400mg ibuprofen and 1000mg Paracetamol at 4 hours in intervals for two days. With a total of 3 doses of ibuprofen and 3 doses of paracetamol per day Then, pain control will be assessed using various primary and secondary outcome scales.

DETAILED DESCRIPTION:
Surgical removal of an impacted mandibular third molar is one of the most common procedures in oral and maxillofacial surgery. Ten million third molars are extracted from approximately 5 million people in the United States each year. Research suggests that wisdom tooth removal has an immediate negative impact on patients' working and social lives: in one study, patients took an average of 1.6 days off work, with over one-third of patients stating that the surgery had affected their performance at work. Postoperative complications may include swelling, bruising, and limited mouth opening, along with difficulty with eating, which can be a major concern to patients and has not been appreciated by healthcare professionals in the past. However, patients are often most concerned about postoperative pain, which may be severe. Approximately one in two patients will experience pain despite analgesic therapy, even one week after surgery. The inflammatory response to surgical trauma is associated with edema, discomfort, dehiscence, and trismus, and these factors may affect the patient's everyday life. The control of these symptoms is frequently based on pharmacological manipulation of local and systemic pain and inflammation mediators. Combining two analgesic agents with distinct mechanisms or sites of action, such as combining a peripherally acting analgesic with a centrally acting analgesic, has been advocated for many years. A common example is the analgesic formulation containing acetaminophen combined with the opioid hydrocodone or paracetamol with ibuprofen. The pain control of single showed that the maximum effect is recorded in the first 2 to 3 hours. Combining two agents tends to increase the effect for 6 to 8 hours. However, as both medication actions commence simultaneously in the latter combination, they are likely to fade in the same way. This may make the patient likely to overdose on such medicine to ensure the continuity of pain relief. This research aims to test the combination of classical pain medication but in a novel alternate way to minimize the dosage and avoid the risk of side effects and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years,
2. Need for surgical extraction of at least one fully or partially impacted lower third molar with a degree of difficulty of 5 points or more on the Pedersen scale,
3. ASA I-II status according to the American Society of Anesthesiologists, and
4. No allergy to the drugs under study.

Exclusion Criteria:

1. Pregnancy
2. Breastfeeding
3. ASA III or above
4. Consumption of antibiotics in the week before surgery; and
5. Clinical evidence of acute infection on the day of surgical intervention
6. Radiographic evidence of peri-radicular pathology in impacted teeth requiring extraction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 48 hours
  Pain was analyzed in 2 ways:
  (1) as the mean of pain intensity VAS score evaluated at 0, 4, 8, 12, 24, 36, and 48 hours post-extraction. Range 0-10
The maximum pain experienced by patients | 48 hours
  a)No pain, b)Some pain, c)Noticeable pain and d)Extreme pain

SECONDARY OUTCOMES:
Onset of pain control | 48 hours
  The time to analgesic onset is defined as the time between trial drug intake and the first report of pain relief,
Duration of pain control | 48 hours
  the time between the first report of perceptible and meaningful pain relief and pain reappearing,
the rescue medicine intake | 48 hours
  the time from trial drug intake to the intake of the first dose of the rescue medicine

CONTACTS AND LOCATIONS:
Overall Officials: Kamis Gaballah, PhD, Principal Investigator — University of Sharjah
Locations (1):
- University dental Hospital, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
The IPD can not be shared

REFERENCES:
- [Background] Friedman JW. The prophylactic extraction of third molars: a public health hazard. Am J Public Health. 2007 Sep;97(9):1554-9. doi: 10.2105/AJPH.2006.100271. Epub 2007 Jul 31. PMID 17666691
- [Background] Colorado-Bonnin M, Valmaseda-Castellon E, Berini-Aytes L, Gay-Escoda C. Quality of life following lower third molar removal. Int J Oral Maxillofac Surg. 2006 Apr;35(4):343-7. doi: 10.1016/j.ijom.2005.08.008. Epub 2005 Nov 8. PMID 16280233
- [Background] Ogden GR, Bissias E, Ruta DA, Ogston S. Quality of life following third molar removal: a patient versus professional perspective. Br Dent J. 1998 Oct 24;185(8):407-10. doi: 10.1038/sj.bdj.4809827. PMID 9828502
- [Background] Savin J, Ogden GR. Third molar surgery--a preliminary report on aspects affecting quality of life in the early postoperative period. Br J Oral Maxillofac Surg. 1997 Aug;35(4):246-53. doi: 10.1016/s0266-4356(97)90042-5. PMID 9291262
- [Background] Kim K, Brar P, Jakubowski J, Kaltman S, Lopez E. The use of corticosteroids and nonsteroidal antiinflammatory medication for the management of pain and inflammation after third molar surgery: a review of the literature. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 May;107(5):630-40. doi: 10.1016/j.tripleo.2008.11.005. Epub 2009 Jan 20. PMID 19157919
- [Background] Mehra P, Reebye U, Nadershah M, Cottrell D. Efficacy of anti-inflammatory drugs in third molar surgery: a randomized clinical trial. Int J Oral Maxillofac Surg. 2013 Jul;42(7):835-42. doi: 10.1016/j.ijom.2013.02.017. Epub 2013 Mar 25. PMID 23535007
- [Background] Hersh EV, Pinto A, Moore PA. Adverse drug interactions involving common prescription and over-the-counter analgesic agents. Clin Ther. 2007;29 Suppl:2477-97. doi: 10.1016/j.clinthera.2007.12.003. PMID 18164916
- [Background] Bailey E, Worthington H, Coulthard P. Ibuprofen and/or paracetamol (acetaminophen) for pain relief after surgical removal of lower wisdom teeth, a Cochrane systematic review. Br Dent J. 2014 Apr;216(8):451-5. doi: 10.1038/sj.bdj.2014.330. PMID 24762895
- [Derived] Gaballah K, Eldohaji T, Tannir ME, Shaban R, Habib R, Ali K. Pain control following impacted mandibular third molar surgery: a comparison of the effectiveness of two different protocols. Sci Rep. 2025 Apr 3;15(1):11519. doi: 10.1038/s41598-025-89744-0. PMID 40181005